CLINICAL TRIAL: NCT03831256
Title: PErsonalized Genomics for Prenatal Abnormalities Screening USing Maternal Blood : Towards First Tier Screening and Beyond
Brief Title: PErsonalized Genomics for Prenatal Abnormalities Screening USing Maternal Blood
Acronym: PEGASUS-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Genome Quebec (Other); Genome British Columbia (Industry); Genome Alberta (Other); Ontario Research Fund (Other); Laval University (Other); St. Justine's Hospital (Other); Ottawa Hospital Research Institute (Other); McGill University (Other); University of British Columbia (Other); University of Alberta (Other); Genome Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, François Rousseau, Professor-doctor, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: SIRUL 118984
Record Dates: First submitted 2019-01-21; First posted 2019-02-05 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Prenatal Disorder; Aneuploidy
Keywords: Real life comparative effectiveness; Non-invasive prenatal screening; Fetal aneuploidy; Randomized controlled trial
MeSH Terms: conditions — Aneuploidy

STUDY DESIGN:
Intervention Model Description: Open-label prospective comparative-effectiveness (utility) randomised trial between first-tier NIPS and the standard of care (2nd-tier NIPS).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (2nd tier NIPS) (Active Comparator): For the standard-of-care arm (2nd tier NIPS) women will undergo Traditional integrated prenatal screening i.e. traditional biochemical (+/- NT) and those with a positive screen for T21 or T18 will be offered Second-tier Non-invasive prenatal screening (NIPS) (for T21, T18, T13) or Invasive prenatal testing for fetal aneuploidy. Ultrasound examination in first and second trimester will be done based on clinical care practice ordered by health care provider. Pregnant women with a positive NIPS test will be offered Invasive prenatal testing for fetal aneuploidy (fetal chromosome analysis).
  Interventions: Diagnostic Test: Traditional integrated prenatal screening; Diagnostic Test: Second-tier Non-invasive prenatal screening (NIPS); Diagnostic Test: Invasive prenatal testing for fetal aneuploidy
- First-tier NIPS (Experimental): For the intervention arm (1st tier NIPS) women will receive First-tier Non-invasive prenatal screening (NIPS) i.e. provide a blood sample between 10-13+5 weeks gestation with NIPS results within 7 - 10 days of sample collection. Ultrasound examination in first and second trimester will be done based on clinical care practice ordered by health care provider. In case of a failed NIPS test (expected to be between 2% and 4% of samples), a new blood sample will be drawn for NIPS retest as well as for a traditional SIPS(serum integrated prenatal screening) or QUAD(quadruple marker prenatal screening) screen (depending on gestational age). Pregnant women with a positive NIPS test will be offered Invasive prenatal testing for fetal aneuploidy (fetal chromosome analysis).
  Interventions: Diagnostic Test: First-tier Non-invasive prenatal screening (NIPS); Diagnostic Test: Invasive prenatal testing for fetal aneuploidy

INTERVENTIONS:
Diagnostic Test: Traditional integrated prenatal screening — biochemical prenatal screening with or without nuchal translucency by US
  Other Names: IPS
  Arms: Standard of care (2nd tier NIPS)
Diagnostic Test: Second-tier Non-invasive prenatal screening (NIPS) — genomics based NIPS after a positive traditional prenatal screen
  Other Names: second tier non-invasive prenatal testing (NIPT)
  Arms: Standard of care (2nd tier NIPS)
Diagnostic Test: First-tier Non-invasive prenatal screening (NIPS) — genomics based NIPS at first trimester
  Other Names: first tier NIPT, Universal NIPS, Universal NIPT
  Arms: First-tier NIPS
Diagnostic Test: Invasive prenatal testing for fetal aneuploidy — amniocentesis or chorionic villi sampling (CVS)

SUMMARY:
This project aims to provide high- quality evidence to inform decisions by health care organisations about using first-tier non-invasive prenatal screening (NIPS) to replace traditional screening tests for trisomy 21, and potentially to screen for other fetal chromosome anomalies. We will compare the current screening approach of second-tier NIPS with the use of first-tier NIPS in a large cohort of pregnant women.

DETAILED DESCRIPTION:
There is some data on the performance of NIPS as a first tier screening test but our systematic review has shown that no trial comparing the effectiveness (utility) of 2nd-tier NIPS with that of first-tier NIPS has been published . Further it is important for health care decision makers to have evidence produced in Canada since the geographical context of healthcare can affect uptake as well as patient decision and thus their healthcare trajectories. There is a need for a trial that is between an explanatory trial and a pragmatic trial to provide the types of answer that we aim to document in the present state of knowledge on NIPS-based screening strategies in Canada. Our Objective is to perform a pan-Canadian large-scale comparative utility (clinical outcomes) study of first-tier NIPS (expanded or not) as compared to the new standard of care (NIPS as a 2nd tier test performed much later during pregnancy and only in high risk pregnancies).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 19 years or older wanting prenatal screening
* 10-13+6 wks determined by dating ultrasound or last menstrual period.
* Not intending to pursue self pay NIPT

Exclusion Criteria:

* Known fetal anomaly at the time of recruitment
* Multiple gestation
* Known twin demise
* Planned CVS or amnio for known genetic condition.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7849 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Gestational age at diagnosis | Up to 24 weeks of gestational age
  gestational age at final result in the sub-set of participants that have received a positive NIPS result and that have been offered diagnostic testing

SECONDARY OUTCOMES:
Gestational age at negative screening result | Up to 24 weeks of gestational age
  gestational age at final result in the sub-set of participants that have received a negative screening result
Gestational age at positive screening result | Up to 24 weeks of gestational age
  gestational age at final result in the sub-set of participants that have received a positive screening result
proportion of women with no results | Up to 24 weeks of gestational age
  proportion of women with no NIPS result at first and second attempt
numbers of days for women with false positive result of screen to wait for result of definite test | Up to 24 weeks of gestational age
  Difference between gestational age (in days) at first positive prenatal screening result and final negative screening result
Change in PROMIS-29 Score | At weeks of gestation 10-13, week 16 and week 22
  The PROMIS-29 assesses seven health domains: physical function, anxiety, depression, fatigue, sleep disturbance, pain interference, and ability to participate in social roles and activities. Each of the seven domains has four questions which are scored on a five-point Likert scale. The PROMIS-29 scales will be scored using a T-score metric method available at the Assessment Center website (http://assessmentcenter.net). A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores mean more of the specific scale's construct, which may indicate a desirable or an undesirable outcome. The assessment will be done at recruitment (10-13 weeks of gestation) and at week 16 and week 22 of gestation.
Change in PROMIS Emotional Distress - Anxiety - Short Form 8a Score | At weeks of gestation 10-13, 16 and 22
  The PROMIS-Anxiety short form assesses anxiety with 8 questions. The form includes 8 items and uses a scale of 1-5 (1=Never, 2=Almost never, 3= Sometimes, 4=Often, 5=Almost always). The raw score is the sum of the points for each response. A higher than average raw score indicates higher than average anxiety. A higher score represents higher levels of anxiety. The assessment will be done at recruitment (10-13 weeks of gestation) and at week 16 and week 22 of gestation.
Patient-Reported Experience Measure (PREM) - Score | At 22 weeks of gestation
  A 17-questions validated PREM questionnaire on pregnancy experience that measures three dimensions - type of prenatal care received and test results (seven questions), pregnancy visits (four questions (scales 1-5) and prenatal screening experience (six questions).
  A profile score by looking at frequencies of responses for each item will be used.
gestational age at termination of pregnancy | Up to 24 weeks of gestational age
  Gestational age at termination of pregnancy for participants having volountary termination
percentage of women undergoing invasive diagnostic testing | Up to 24 weeks of gestational age
  see outcome title

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Langlois, MD FRCPC, Principal Investigator — University of British Columbia; Francois Rousseau, MD MSc FRCPC, Principal Investigator — CHU de Québec - Université Laval
Locations (6):
- Canada (6):
  - Kelowna Regional Fertility Center, Kelowna, British Columbia
  - Prince Rupert Regional Hospital, Prince Rupert, British Columbia
  - Children's & Women's Health Centre, Vancouver, British Columbia
  - CHU Ste-Justine, Montreal, Quebec
  - CHU de Québec - Université Laval, Québec, Quebec
  - CIUSSS Côte-Nord, Sept-Îles, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Badeau M, Lindsay C, Blais J, Nshimyumukiza L, Takwoingi Y, Langlois S, Legare F, Giguere Y, Turgeon AF, Witteman W, Rousseau F. Genomics-based non-invasive prenatal testing for detection of fetal chromosomal aneuploidy in pregnant women. Cochrane Database Syst Rev. 2017 Nov 10;11(11):CD011767. doi: 10.1002/14651858.CD011767.pub2. PMID 29125628